CLINICAL TRIAL: NCT02583607
Title: Brava and Fat Transfer for Breast Reconstruction
Acronym: Brava
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Yoav Gronovich, Certified Plastic Surgeon, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81/15
Record Dates: First submitted 2015-10-14; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Fat Necrosis of Breast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brava and fat transfer (Experimental): The purpose of the study is to examine the efficacy of Brava with fat grafting in woman undergoing mastectomy in the institution.
  Woman who will agree to participate in the study will be instructed how to wear the Brava, and after 200 hours of using the device they will be operated for fat transfer to the breast in order to reconstruct it.
  Interventions: Device: Brava

INTERVENTIONS:
Device: Brava — The purpose of the study is to examine the efficacy of Brava with fat grafting in woman undergoing mastectomy in the institution.
  woman who will agree to participate in the study will be instructed how to wear the Brava, and after 200 hours of using the device they will be operated for fat transfer to the breast in order to reconstruct it.

SUMMARY:
Breast reconstruction is one of the most challenging aspects in plastic surgery. One of the most sophisticated methods of breast reconstruction is using of autologous fat grafting. Brava is a device that invented by Dr Roger Khouri, and is intended to improve the final results of fat grafting.

DETAILED DESCRIPTION:
The purpose of the study is to examine the efficacy of Brava with fat grafting in woman undergoing mastectomy in the institution. Woman who will agree to participate in the study will be instructed how to wear the Brava, and after 200 hours of using the device they will be operated for fat transfer to the breast in order to reconstruct it.

ELIGIBILITY:
Inclusion Criteria:

* woman after mastectomy

Exclusion Criteria:

* smokers
* collagen disease
* low compliance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients satisfied with breast reconstruction using Brava and fat transfer | 6 months
  patients undergoing breast mastectomy will undergo breast reconstruction using the Brava and fat transfer, and will be assessed by a certified plastic surgeon who will not be a part of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Gronovich, MD, Study Director — Shaare Zedek Medical Center

REFERENCES:
- See also: The BRAVA Breast Enhancement and Shaping System — http://brava.com/